CLINICAL TRIAL: NCT02678117
Title: Analgesic Potentials of Preoperative Oral Pregabalin,Intravenous Magnesium Sulphate and Their Combination in Acute Post-thoracotomy Pain.(Randomized,Double-Blind Study)
Brief Title: Analgesic Potentials of Preoperative Pregabalin,Magnesium Sulphate and Their Combination in Acute Post-thoracotomy Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Salah Ahmed Abd Elgalil, Demonstrator in anaesthesia department, National Cancer Institute, Egypt, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI,IRB 2010014053.3
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pregabalin & placebo (Active Comparator): : will receive single dose oral Pregabalin 300 mg one hour preoperative and 200 ml of normal saline over 20 min.
  Interventions: Drug: Pregabalin & Placebo
- Magnesium sulphate & Placebo (Active Comparator): will receive preoperative single dose IV Magnesium Sulphate 50mg /kg infused over 20 minutes diluted in 200 ml normal saline and a placebo capsule similar to pregabalin 300 mg.
  Interventions: Drug: Magnesium sulphate & Placebo
- Pregabalin & Magnesium sulphate (Active Comparator): : will receive single dose oral pregabalin 300mg one hour preoperative and single dose IV Magnesium Sulphate 50mg /kg infused over 20 minutes diluted in 200 ml normal saline.
  Interventions: Drug: Pregabalin & Magnesium sulphate
- Placebo (Placebo Comparator): will receive placebo medications at the same time and route of administration of other groups.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin & Placebo
  Arms: Pregabalin & placebo
Drug: Magnesium sulphate & Placebo
  Arms: Magnesium sulphate & Placebo
Drug: Pregabalin & Magnesium sulphate
  Arms: Pregabalin & Magnesium sulphate
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study evaluates the effect of giving preoperative adjuvant drug as pregabalin or magnesium sulphate or a combination of both drugs to decrease postoperative morphine consumption and pain intensity in the first 24 hours in postoperative period . quarter of patients receive single dose oral pregabalin 300mg 1 hour preoperatively ,other quarter receive single intravenous Magnesium sulphate 50mg per Kg over 200ml saline over 20 minutes preoperatively , other quarter receive combination of both drugs , the last quarter receive placebo drugs . All patients receive 0.1mg per Kg intravenous morphine sulphate intraoperatively

DETAILED DESCRIPTION:
Magnesium (Mg) acts on N-methyl-D-aspartate (NMDA) receptor as a non-competitive antagonist with antinociceptive effects.

Gabapentin is an alkylated analogue of gammaaminobutyric acid (GABA) developed primarily as an anticonvulsant drug. It was described as an analgesic drug for the treatment of neuropathic pain in the 1990s. Although it is named Gabapentin,it does not bind at the GABA A or GABA B receptor. It binds with high affinity for the α2δ subunit of the presynaptic voltage-gated calcium channels, which reduce calcium-dependent release of pro-nociceptive neurotransmitters in the pain pathways. Pregabalin is a structural analogue of GABA was introduced after Gabapentin. If we used these drugs in combination to opioids preoperatively as preventive analgesia may decrease postoperative opioid consumption and pain intensity.

ELIGIBILITY:
Inclusion Criteria:

1. ASA status of1 or 2
2. Patients undergoing thoracotomy
3. Body mass index (BMI): Less than forty and more than twenty.

Exclusion Criteria:

- 1. Known sensitivity or contraindication to drugs used in the study. 2. History of psychological disorders and/or chronic pain. 3. Patients receiving medical therapies that are considered to result in tolerance to opioids.

4. Significant liver or kidney diseases that will affects the pharmacokinetics of study drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | First 24 hours in postoperative period
  patients are given regular intravenous morphine through patient controlled analgesia (PCA) and morphine consumption calculated from the PCA device

SECONDARY OUTCOMES:
Pain intensity using Visual Analogue Scale | First 24 hours in postoperative period
  Assessment of pain intensity every 4 hours in the first 24 hours in postoperative period
Recovery Time | Immediately after ending the surgery
  Time taken for recovery of the patient to be fully awake
Heart Rate | First 24 hours in postoperative period
  Assessment of Heart Rate every 4 hours
Blood Pressure | First 24 hours in postoperative period
  Assessment of Blood Pressure every 4 hours
Oxygen saturation | First 24 hours in postoperative period
  Assessment of Oxygen saturation every 4 hours
Respiratory Rate | First 24 hours in postoperative period
  Assessment of Respiratory Rate every 4 hours
Postoperative nausea and vomiting | First 24 hours in postoperative period
  Postoperative nausea and vomiting scale (none 0, mild 1, moderate 2 , sever 3)
Side effects from the used drugs | First 24 hours in postoperative period
Sedation score | First 24 hours in postoperative period
  Using Ramsay Sedation score

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa A Ahmed, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be available within 6 months of study completion

REFERENCES:
- [Background] Sagit M, Yalcin S, Polat H, Korkmaz F, Cetinkaya S, Somdas MA. Efficacy of a single preoperative dose of pregabalin for postoperative pain after septoplasty. J Craniofac Surg. 2013 Mar;24(2):373-5. doi: 10.1097/SCS.0b013e31827fece5. PMID 23524696
- [Background] Kiran S, Gupta R, Verma D. Evaluation of a single-dose of intravenous magnesium sulphate for prevention of postoperative pain after inguinal surgery. Indian J Anaesth. 2011 Jan;55(1):31-5. doi: 10.4103/0019-5049.76605. PMID 21431050
- [Derived] Salah Abdelgalil A, Shoukry AA, Kamel MA, Heikal AMY, Ahmed NA. Analgesic Potentials of Preoperative Oral Pregabalin, Intravenous Magnesium Sulfate, and their Combination in Acute Postthoracotomy Pain. Clin J Pain. 2019 Mar;35(3):247-251. doi: 10.1097/AJP.0000000000000673. PMID 30730476